CLINICAL TRIAL: NCT03536065
Title: Post-Discharge Opioid Reduction Intervention for Open, Laparoscopic, and Endoscopic Surgery (ORIOLES): A Quality Improvement Study of Prescribing Habits and Patient Education
Brief Title: Post-Discharge Opioid Reduction Intervention for Open, Laparoscopic, and Endoscopic Surgery
Acronym: ORIOLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00162359
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer; Opioid Use
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Pre-Post Study Design with Non-Pharmacologic Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Intervention (Active Comparator): Current practice (unchanged)
  Interventions: Behavioral: Current Care
- Post-Intervention (Experimental): Reduction of opioid prescription based on Pre-Intervention data, implementation of a discharge sheet and nursing education.
  Interventions: Behavioral: Opioid Reduction Intervention

INTERVENTIONS:
Behavioral: Opioid Reduction Intervention — Patient education discharge sheet, nursing education, opioid prescription reduction based on Pre-Intervention data
  Arms: Post-Intervention
Behavioral: Current Care — Current unchanged care provided; unchanged provider prescribing and unchanged education of patients prior to intervention
  Arms: Pre-Intervention

SUMMARY:
ORIOLES is a non-randomized, pre-post intervention study designed to improve quality of opioid prescribing and use after discharge for patients undergoing urologic surgery. The study will initially focus on a pre-defined cohort of patients undergoing radical prostatectomy. After the predefined study period for the pre-intervention arm, a three-part intervention is employed to assess the effect on opioid prescribing and use in the post-intervention arm. Pending results, the intervention may be applied to all surgeries in the department for routine clinical care.

DETAILED DESCRIPTION:
The goal of the study is to reduce the amount of opioid analgesia prescribed after urologic surgery in the Department of Urology at Johns Hopkins. The initiative focuses on patients undergoing surgery for prostate cancer with radical prostatectomy including patients enrolled in IRB00123618/NCT03006562. The pre-intervention arm will consist of patients enrolled August 2017 to January 2018. The intervention arm will consist of patient enrolled January 2018 to completion of the study.

The intervention consists of a information discharge sheet, a standardized prescribing guideline at discharge, and nurses providing improved education for patients at discharge about appropriate use of opioid medication, routes for disposal, and potential side effects. Data on prescriptions written (amount and type of mediation) and use of opioid and other pain medication after surgery will be compared before and after the quality improvement initiative is started. Outcomes are assessed via 30-day phone call follow-up with data on perioperative outcomes, postoperative medication use, and symptoms already assessed in IRB00123618/NCT03006562. At the completion of the pre-intervention arm, providers in the urology department are informed about the average and distribution of usage of post-discharge opioids. Education and standardized prescribing (allowing for provider judgment) may help reduce/personalize the amount of opioids prescribed at discharge to reduce wasted medication entering circulation. The initiative may then be expanded to encompass all surgeries in the department to reduce opioid prescribing and use for routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with prostate cancer and enrolled in NCT03006562

Exclusion Criteria:

* Patients not undergoing radical prostatectomy (for the primary pre-post ORIOLES study)

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Opioid Use | 30 days
  The total oral morphine equivalents (OMEQ) used by the patient up to 30 days after discharge from the hospital

SECONDARY OUTCOMES:
Opioid Prescription | Discharge date
  The total oral morphine equivalents (OMEQ) prescribed by the inpatient provider to the patient at discharge after surgery
Opioid Disposal | 30 days
  Method of disposal (if any) by the patient of opioid medication prescribed for post-discharge use
Need for Refill or Additional Opioid Medication | 30 days
  Patient obtaining any additional opioid medication for post-surgical pain within 30 days after discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Amin S Herati, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang MM, Su ZT, Becker REN, Pavlovich CP, Partin AW, Allaf ME, Patel HD. Complications after open and robot-assisted radical prostatectomy and association with postoperative opioid use: an analysis of data from the PREVENTER trial. BJU Int. 2021 Feb;127(2):190-197. doi: 10.1111/bju.15172. Epub 2020 Aug 17. PMID 32654363
- [Result] Patel HD, Srivastava A, Patel ND, Faisal FA, Ludwig W, Joice GA, Schwen ZR, Allaf ME, Han M, Herati AS. A Prospective Cohort Study of Postdischarge Opioid Practices After Radical Prostatectomy: The ORIOLES Initiative. Eur Urol. 2019 Feb;75(2):215-218. doi: 10.1016/j.eururo.2018.10.013. Epub 2018 Oct 21. PMID 30352714
- [Result] Patel HD, Faisal FA, Patel ND, Pavlovich CP, Allaf ME, Han M, Herati AS. Effect of a prospective opioid reduction intervention on opioid prescribing and use after radical prostatectomy: results of the Opioid Reduction Intervention for Open, Laparoscopic, and Endoscopic Surgery (ORIOLES) Initiative. BJU Int. 2020 Mar;125(3):426-432. doi: 10.1111/bju.14932. Epub 2019 Nov 15. PMID 31643128